CLINICAL TRIAL: NCT02870894
Title: Electrical Impedance Tomography for Quantification of Pulmonary Edema in Acute Respiratory Distress Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, He Hongli, Principal Investigator, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH
Record Dates: First submitted 2016-08-14; First posted 2016-08-17 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Evaluation of pulmonary edema is a key factor in monitoring and guidance of therapy in acute respiratory distress syndrome (ARDS) patients. To date, methods available at the bedside for estimating the physiologic correlate of pulmonary edema, extravascular lung water(EVLW), often are unreliable or require invasive measurements. The purpose of the this study is to develop a novel approach to reliably assess extravascular lung water by electrical impedance tomography(EIT).

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in this study if the following criteria have been met:

1. Males and females > 18 years old and <85 years old (non-pregnant, non-lactating females).
2. Patients fulfilled the Berlin diagnostic criteria of ARDS
3. Signed written informed consent has been obtained
4. Patients had monitoring system Pulse-Induced Contour Cardiac Output (PiCCO)

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Patients with contraindication of EIT(Skin abrasions or wounds in the chest area.Patients with pacemakers or paced EKG rhythms.Thoracic deformity. Severe subcutaneous emphysema)
3. Patients <18 years old or > 85 years old
4. Patients Without monitoring system Pulse-Induced Contour Cardiac Output (PiCCO)
5. Patients with Cardiac function of grade 4 or patients with acute myocardial infarction or acute coronary syndrome

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients with ARDS will be enrolled between August 2016 and August 2017 when they fulfilled the inclusion criteria,and unfulfilled the exclusion criteria below
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Comparison between a novel EIT-based method to estimate pulmonary edema (lung water ratio-EIT ) with a conventional measurement for EVLW using trans-cardiopulmonary thermodilution technique | once the patient was consented and enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Huang, MD, Principal Investigator — Sichuan Academy of Medical Sciences
Locations (1):
- Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhao Z, He H, Luo J, Adler A, Zhang X, Liu R, Lan Y, Lu S, Luo X, Lei Y, Frerichs I, Huang X, Moller K. Detection of pulmonary oedema by electrical impedance tomography: validation of previously proposed approaches in a clinical setting. Physiol Meas. 2019 Jun 4;40(5):054008. doi: 10.1088/1361-6579/ab1d90. PMID 31035265